CLINICAL TRIAL: NCT01417975
Title: Does an Acute Bout of Exercise Affect Smoking Satisfaction?
Brief Title: Effect of an Acute Bout of Exercise on Smoking Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SmokingTopography1114
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2012-06

CONDITIONS: Cancer
Keywords: exercise; smoking satisfaction; topography; cravings
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Exercise Group (Experimental): The moderate exercise condition will involve participants waking briskly (equivalent to moderate intensity) on a treadmill for 10 minutes. Moderate intensity exercise is defined as 40-68% of heart rate reserve (HRR). Heart rate (HR) will be monitored using a Polar RS100 Heart Rate monitor to serve as a guide for participants to attain the appropriate intensity.
  Interventions: Behavioral: Moderate Exercise Group
- Passive Sitting Group (Active Comparator): The passive sitting condition will involve participants sitting passively in a chair for 10 minutes. Heart rate (HR) will be monitored in participants of the passive sitting group to help maintain group equivalency (with the moderate exercise condition) with regards to distraction effects and researcher contact.
  Interventions: Behavioral: Passive Sitting Group

INTERVENTIONS:
Behavioral: Moderate Exercise Group — Participants will be required to walk briskly (equivalent to moderate intensity) on a treadmill for 10 minutes.
  Other Names: Physical activity
  Arms: Moderate Exercise Group
Behavioral: Passive Sitting Group — Participants will be required to sit passively on a chair for 10 minutes.
  Other Names: Sedentary
  Arms: Passive Sitting Group

SUMMARY:
Female and male smokers will complete questionnaires and smoking behavior will be examined. After abstaining from smoking for approximately 18 hours, they will be randomized to a moderate intensity exercise groups or passive sitting group. Smoking satisfaction and smoking behavior will be assessed following treatment.

The hypotheses detailed below are specific to the randomization of participants into the following 2 groups:

1. Moderate exercise (Experimental condition; MEG)
2. Passive sitting (Attention control condition; PSG)

Hypothesis 1: A bout of moderate intensity exercise will be associated with decreased smoking satisfaction after a temporary period of abstinence compared to a control condition.

Hypothesis 2: Smoking topographic measures will mediate the relationship between a bout of moderate intensity exercise and smoking satisfaction.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in Canadians (Canadian Cancer Society (CCS), 2010). Cigarette smoking is responsible for 85% of these cases (CCS, 2007). Exercise has been shown to be an effective adjunct to pharmacological cessation strategies (Ussher, Taylor, & Faulkner, 2008). A recent systematic review concluded that a single bout of low to moderate intensity exercise can help regulate cravings, withdrawal symptoms and negative affect associated with quitting (Taylor, Ussher, & Faulkner, 2007).

Smoking satisfaction is an immediately reinforcing effect of nicotine. Smoking satisfaction may outweigh the temporally distant adverse health risks of smoking (Cappelleri, Bushmakin, Baker, Merikle, Olufade, & Gilbert, 2007). Varenicline, an alpha 4-beta-2 nAChR partial agonist, mimics the effect of nicotine by reducing cravings and withdrawal symptoms (Coe et al., 2005). A 12-week treatment period of varenicline has been shown to reduce smoking satisfaction (Jorenby et al., 2006). However, the effect of acute exercise on smoking satisfaction is not yet known.

Smoking topography is a key facet of smoking behaviour. Smoking behaviour can be subjectively or objectively measured by quantifying puff volume, maximum puff velocity, inter-puff interval, puff duration, number of puffs per cigarette and time to smoke a single cigarette. Smoking topography can estimate exposure to carcinogenic toxins present in cigarette smoking (Djordjevic, Hoffman, & Hoffman, 1997). Evidence exists to support that exercise modifies smoking topography (Katomeri & Taylor 2006; Mikhail, 1983; Reeser, 1983; Zacny & Stitzer, 1985).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age
* Smoke 10 or more cigarettes per day
* Not have any medical condition that is contraindicative for exercise
* Not be pregnant or intending on becoming pregnant over the course of the study
* Be able to read and write in English
* Have a telephone or e-mail account so they can be contacted
* Successful completion of the Physical Activity Readiness Questionnaire (PAR-Q)
* Have a Medical Doctor's clearance if they answer "YES" to one or more questions on the Physical Activity Readiness Questionnaire (PAR-Q)
* Have not been engaged in a serious quit attempt in the last six months
* Have been smoking for more than 2 years
* Must not be suffering from an illness (e.g. cold) that would affect their typical smoking behaviour

Exclusion Criteria:

* Contraindication to exercise (e.g. disability, unstable angina)
* On medication for physical and/or mental health reasons that would make compliance with the study protocol difficult or dangerous
* Have substance dependency problems (e.g. alcohol)
* Are pregnant
* Be younger than 18 years of age
* Be 64 years or older prior to completion of the study
* Have been engaged in a serious quite attempt in the last six months
* Have been smoking for less than 2 years
* Suffering from an illness (e.g. cold) that would affect their typical smoking behaviour

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Smoking satisfaction | One week
  Smoking satisfaction will be assessed using the 12-item modified version of the Cigarette Evaluation Questionnaire (mCEQ; Cappelleri, Bushmakin, Baker, Merikle, Olufade & Gilbert, 2007).

SECONDARY OUTCOMES:
Smoking topography | One week
  Smoking topography will be assessed using the Clinical Research Support System (CReSS) Pocket, a computer-based, battery-powered, hand-held unit by Plowshare Technologies. The CReSS Pocket has an orifice flow meter mouthpiece, and a pressure drop related to the flow rate that is produced when a puff is taken. From the flow rate, the CReSS derives puff count (number of puffs per cigarette), puff volume (the volume of carbon monoxide taken in during each puff), puff duration (length of time for each puff), inter-puff interval (amount of time between puffs), and time to first puff.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — The University of Western Ontario
Locations (1):
- The Exercise and Health Psychology Laboratory - The University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Ussher MH, Taylor A, Faulkner G. Exercise interventions for smoking cessation. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD002295. doi: 10.1002/14651858.CD002295.pub3. PMID 18843632
- [Background] Taylor AH, Ussher MH, Faulkner G. The acute effects of exercise on cigarette cravings, withdrawal symptoms, affect and smoking behaviour: a systematic review. Addiction. 2007 Apr;102(4):534-43. doi: 10.1111/j.1360-0443.2006.01739.x. PMID 17286639
- [Background] Taylor A, Katomeri M. Walking reduces cue-elicited cigarette cravings and withdrawal symptoms, and delays ad libitum smoking. Nicotine Tob Res. 2007 Nov;9(11):1183-90. doi: 10.1080/14622200701648896. PMID 17978993
- [Background] West R, Baker CL, Cappelleri JC, Bushmakin AG. Effect of varenicline and bupropion SR on craving, nicotine withdrawal symptoms, and rewarding effects of smoking during a quit attempt. Psychopharmacology (Berl). 2008 Apr;197(3):371-7. doi: 10.1007/s00213-007-1041-3. Epub 2007 Dec 15. PMID 18084743
- See also: Exercise and Health Psychology Laboratory — http://www.ehpl.uwo.ca